CLINICAL TRIAL: NCT02002156
Title: A Pilot Study of the Impact of BCG Administration on the Immunogenicity of Serogroup C Meningococcal Conjugate Vaccine in Healthy Infants
Brief Title: A Study of the Interaction Between BCG And MenC Immunisation: BAM
Acronym: BAM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OVG-2013/04
Record Dates: First submitted 2013-11-19; First posted 2013-12-05 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: BCG Infection; Reaction - Vaccine; Immune Response
MeSH Terms: interventions — diphtheria-tetanus-five component acellular pertussis-inactivated poliomyelitis -Haemophilus influenzae type b conjugate vaccine; Diphtheria-Tetanus-acellular Pertussis Vaccines; 13-valent pneumococcal vaccine; Measles-Mumps-Rubella Vaccine; RIX4414 vaccine; BCG Vaccine; halofantrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- BCG at birth and routine vaccines (Experimental): BCG, NeisVac-C®, Pediacel®, Infanrix™, Prevenar-13®, Menitorix®, Priorix®, Rotarix®
  Interventions: Biological: BCG, NeisVac-C®, Pediacel®, Infanrix™, Prevenar-13®, Menitorix®, Priorix®, Rotarix®
- BCG at 3 months old and routine vaccines (Experimental): BCG, NeisVac-C®, Pediacel®, Infanrix™, Prevenar-13®, Menitorix®, Priorix®, Rotarix®
  Interventions: Biological: BCG, NeisVac-C®, Pediacel®, Infanrix™, Prevenar-13®, Menitorix®, Priorix®, Rotarix®
- Routine vaccines (Experimental): NeisVac-C®, Pediacel®, Infanrix™, Prevenar-13®, Menitorix®, Priorix®, Rotarix®
  Interventions: Biological: NeisVac-C®, Pediacel®, Infanrix™, Prevenar-13®, Menitorix®, Priorix®, Rotarix®

INTERVENTIONS:
Biological: BCG, NeisVac-C®, Pediacel®, Infanrix™, Prevenar-13®, Menitorix®, Priorix®, Rotarix® — This group will receive BCG at birth and all routine vaccinations.
  Other Names: BCG vaccine (Serum Statens Institute); NeisVac---C®, Baxter Healthcare Ltd.; Pediacel®, Sanofi Pasteur MSD Ltd.; Infanrix™---IPV---Hib, GlaxoSmithKline; Prevenar---13®, Pfizer Ltd.; Menitorix®, GlaxoSmithKline UK; Priorix®, GlaxoSmithKline UK; Rotarix®, GlaxoSmithKline UK
  Arms: BCG at birth and routine vaccines
Biological: BCG, NeisVac-C®, Pediacel®, Infanrix™, Prevenar-13®, Menitorix®, Priorix®, Rotarix® — This group will receive BCG at three months old and all routine vaccinations.
  Other Names: BCG vaccine (Serum Statens Institute); NeisVac---C®, Baxter Healthcare Ltd.; Pediacel®, Sanofi Pasteur MSD Ltd.; Infanrix™---IPV---Hib, GlaxoSmithKline; Prevenar---13®, Pfizer Ltd.; Menitorix®, GlaxoSmithKline UK; Priorix®, GlaxoSmithKline UK; Rotarix®, GlaxoSmithKline UK
  Arms: BCG at 3 months old and routine vaccines
Biological: NeisVac-C®, Pediacel®, Infanrix™, Prevenar-13®, Menitorix®, Priorix®, Rotarix® — This group will receive no BCG but will receive all routine vaccinations.
  Other Names: NeisVac---C®, Baxter Healthcare Ltd.; Pediacel®, Sanofi Pasteur MSD Ltd.; Infanrix™---IPV---Hib, GlaxoSmithKline; Prevenar---13®, Pfizer Ltd.; Menitorix®, GlaxoSmithKline UK; Priorix®, GlaxoSmithKline UK; Rotarix®, GlaxoSmithKline UK
  Arms: Routine vaccines

SUMMARY:
The Bacille Calmette-Guérin (BCG) vaccine is the only vaccine licenced to prevent tuberculosis (TB). The stimulus it gives to the immune system allows it to respond more effectively to a subsequent infection with TB.

Many studies have shown that BCG is effective in reducing deaths from TB disease, particularly in children. However, there is also evidence that in countries with a relatively high death rate, BCG reduces this death rate but by more than would be expected by its effect on TB alone. This controversial but important finding warrants further and serious consideration. One possibility is that BCG, in addition to stimulating the immune system against TB, also has a positive effect on the way the immune system works more generally. This might mean a more effective response to serious infections that are completely unrelated to TB, or the ability to respond better to other routine childhood vaccines, or to maintain such responses for longer. In these examples, the timing of BCG administration in relation to other vaccines could be crucial.

This study will recruit 30 healthy babies who would not routinely be offered the BCG vaccine in the UK within the first week of life. Babies will be assigned at random to one of three groups of ten babies each. BCG will be given to one group of babies around birth, one at three months old and the last group will not get BCG during the study. Babies will stay in the study until 13 months old and have five blood tests over this period.

This preliminary study will look at the participants' blood to see if there are differences in the immune system, or its response to the MenC childhood meningitis vaccine or the pattern of genes activated after BCG has been given.

ELIGIBILITY:
Inclusion Criteria:

Healthy male or female babies aged 7 days or under

* Born at term (≥ 36 completed weeks of gestation)
* Valid informed consent provided by an individual with parental responsibility (parent or legal guardian)
* Living within the Thames Valley region at enrolment without intention to move out of this region during the course of the study
* Parents or legal guardians must be aged 18 years or over
* Parent or legal guardian is able (in the Investigator's opinion) and willing to comply with all study requirements
* Parent or legal guardian consent provided for General Practitioner and consultant, if appropriate, to be notified of participation in the study
* Parent or legal guardian consent to review hospital birth records before enrolment and inform GP or Consultant of involvement in study, if appropriate

Exclusion Criteria:

Confirmed, suspected or significant risk of immunodeficiency (including but not limited to: maternal history of Human Immunodeficiency Virus infection, family history of congenital or hereditary immunodeficiency and receipt of significant immunosuppressive medication by the participant during the study, or by the mother prior to delivery)

* Receipt of BCG or another live vaccine prior to enrolment
* Receipt of any vaccine, either prior to enrolment or planned during the study, except for:

  * those listed in the study protocol at the times indicated
  * hepatitis A or B vaccine or influenza vaccine.
* Receipt prior to enrolment, or planned receipt during the study, of monoclonal antibodies, immunoglobulin or any blood product
* A baby who would normally be offered BCG at birth under current Department of Health guidance3. This means:

  * babies living in an area of the UK with an annual incidence of TB >40 / 100,000 or
  * babies who have a parent or grandparent who was born in a country with an annual incidence of TB >40 / 100,000
* Confirmed or suspected household contact with active TB
* Confirmed or suspected anaphylaxis to any component of BCG or other study vaccine
* Any confirmed or suspected serious medical condition (including seizures, neurological conditions, major congenital abnormalities or malignancy)
* Receipt of systemic antimicrobial medication since birth
* Parents or legal guardians should not be members of the study team or named on the study delegation log
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the potential participant (or carer) at risk because of participation in the study, or may influence the result of the study, or the potential participant's ability to participate in the study.
* A potential participant who has participated or is participating in another research study involving an investigational product

Max Age: 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2014-06-20 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2018-06-27 (Actual)

PRIMARY OUTCOMES:
MenC-specific IgG in blood | 8 weeks following the dose of MenC vaccine (i.e. at 20 weeks of age if no delay in the schedule)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oxford, Oxford Vaccine Group, Oxford, Oxfordshire, United Kingdom